CLINICAL TRIAL: NCT01366261
Title: Rigid Versus Semirigid Thoracoscopy in Diagnosing Pleural Diseases: a Randomized Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aleš Rozman (Other)
Responsible Party: Sponsor-Investigator, Aleš Rozman, MD, The University Clinic of Pulmonary and Allergic Diseases Golnik
Organization: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: endo-0001
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Pleural Diseases
Keywords: Flex-rigid pleuroscopy; pleural biopsy; pleural effusion; safety; thoracoscopy
MeSH Terms: conditions — Pleural Diseases; Pleural Effusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- semirigid thoracoscopy (Experimental): Semirigid instrument which we compare was autoclavable Olympus LTF-160 (Olympus Tokyo, Japan). Handle and its controls were similar to flexible fiberoptic bronchoscope, with the insertion portion composed of 22 cm long rigid part and distal 5 cm flexible tip with angulation range 1600 up / 1300 down. The external diameter of insertion portion was 7 mm with 2,8 mm inner channel diameter. The instrument was compatible with Olympus EVIS Exera 160 and 145 and EVIS 100 and 140 video processors and light sources, otherwise employed in video-bronchoscopy. Forceps, which we used was flexible FB-55CD-1 Olympus forceps with 5 mm long cusps and diameter, which fitted the diameter of inner channel of semirigid thoracoscope.
  Interventions: Device: semirigid thoracoscopy
- rigid thoracoscopy (Active Comparator): The rigid instrument was autoclavable OP EndoEYE WA50120A (Olympus Tokyo, Japan) video thoracoscope. The length of the instrument was 29 cm with 00 direction of view and 700 field of view. The external diameter of the instrument was 10 mm with 5,2 mm inner channel diameter. The instrument was compatible with Olympus Visera OTV-S7V and EVIS Exera II CV-180 video processors. Cusps of rigid forceps had outer diameter 5 mm and length 10 mm.
  Interventions: Device: rigid thoracoscopy

INTERVENTIONS:
Device: semirigid thoracoscopy — thoracoscopy with semirigid instrument
  Other Names: autoclavable Olympus LTF-160 (Olympus Tokyo, Japan)
  Arms: semirigid thoracoscopy
Device: rigid thoracoscopy — thoracoscopy with rigid instrument
  Other Names: autoclavable OP EndoEYE WA50120A (Olympus Tokyo, Japan) video thoracoscope
  Arms: rigid thoracoscopy

SUMMARY:
The purpose of our study was to compare the size and the quality of biopsy samples together with the diagnostic adequacy of semirigid thoracoscopy with that of rigid instrument in prospective, randomized fashion. The second aim was to compare safety and tolerability of both types of procedure, performed in local anesthesia with addition of intravenous sedation and analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 18 or more years old
* unilateral pleural effusion of unknown origin
* pleural irregularities suspicious for pleural malignancy
* referral for thoracoscopy after less invasive means of diagnosis had failed

Exclusion Criteria:

* uncontrolled bleeding tendency
* unstable cardiovascular status
* severe heart failure
* ECOG performance status 4
* persistent hypoxemia after evacuation of pleural fluid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
diagnostic adequacy of semirigid thoracoscopy | 12 months
  * comparison of diagnostic adequacy of both instruments (number of definitive diagnosis in each group)
  * size of the biopsy specimens in mm2
  * interpretability of biopsy specimens in histopathology terms: 1. easily interpretable (enough tissue with all elements required for diagnosis) 2. interpretable with some difficulty (less tissue or diagnostic elements - diagnosis less reliable) 3. interpretable with great difficulty (little tissue or scarce diagnostic elements - low reliability of diagnosis) 4. non-interpretable (diagnosis not possible)

SECONDARY OUTCOMES:
safety | 1 month
  Major adverse events:
  * bleeding
  * infection
  * reexpansion pulmonary edema
  Minor adverse events:
  * transient self-limited fever
  * pain
  * prolongued air leak
  * subcutaneous emphysema
    30-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic Golnik, Golnik, Golnik, Slovenia

REFERENCES:
- [Derived] Rozman A, Camlek L, Marc-Malovrh M, Triller N, Kern I. Rigid versus semi-rigid thoracoscopy for the diagnosis of pleural disease: a randomized pilot study. Respirology. 2013 May;18(4):704-10. doi: 10.1111/resp.12066. PMID 23418922